CLINICAL TRIAL: NCT04810884
Title: Fractures and Bone Disease in Living Kidney Donors
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Rajiv Kumar, M.D., Principal Investigator, Mayo Clinic
Other Study IDs: 20-004432; R01DK125252 (NIH)
Record Dates: First submitted 2021-02-15; First posted 2021-03-23 (Actual); Last update posted 2023-10-11 (Actual); Status verified 2023-10

CONDITIONS: Renal Transplant Donor of Left Kidney; Renal Transplant Donor of Right Kidney

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Living kidney donors: Aim 1: A survey about fractures and general bone health will be sent to 3000 prior living kidney donors.
  Aim 2: Out of these 3000 subjects, 200 prior living kidney donors who are ≥10 years post kidney donation will be invited to Mayo Clinic Rochester for an assessment of bone health. Each subject will undergo lateral DXA with vertebral fracture assessment (VFA), bone density assessment of each hip, radius and spine by DXA scan, bone structure assessment by HRpQCT of the distal radius and tibia, finite element assessment (µFEA), skin AGEs measurement, and blood collection to measure markers of bone formation and resorption.
- Matched Controls: Aim 1: A survey about fractures and general bone health will be sent to 3000 age, sex, race, and comorbidity-matched subjects who would have been eligible to donate but did not donate a kidney.
  Aim 2: Out of these 3000 subjects, 200 control subjects who would be eligible to donate, but have not donated, and are matched by age, sex, race, and comorbidity to donors at the time of donation will be invited to Mayo Clinic Rochester for an assessment of bone health. Each subject will undergo lateral DXA with vertebral fracture assessment (VFA), bone density assessment of each hip, radius and spine by DXA scan, bone structure assessment by HRpQCT of the distal radius and tibia, finite element assessment (µFEA), skin AGEs measurement, and blood collection to measure markers of bone formation and resorption.

SUMMARY:
This research study is being done to measure bone health in living kidney donors and compare them to non-kidney donors to learn if living kidney donors have a higher risk of bone fractures (breaks) after kidney donation. Certain chemicals in the body that help maintain bone health were shown to have changed after kidney donation in living donors, whether or not these changes lead to a decrease in bone quality and increase the risk of fractures is not known.

The purpose of this study is to compare the bone health of living kidney donors, with the bone health of non-kidney donors. This information will be helpful in informing future kidney donors of the risks of donation and in creating treatments to help prevent these complications.

DETAILED DESCRIPTION:
This is an observational study that consists of two Aims:

Aim 1 is a survey sent to 3000 prior living kidney donors and 3000 matched controls. The survey contains questions about history of bone fractures and general bone health. Prior living kidney donors will be identified and surveyed from three Minnesota centers: Mayo Clinic, Rochester; Hennepin County Medical Center (HCMC); and the University of Minnesota (UMN).

Aim 2 of this study includes an assessment of bone structure and bone turnover markers in a subset of donors and matched controls. 200 prior living kidney donors and 200 matched controls will be invited to Mayo Clinic Rochester's CRTU for an assessment of bone health. Each subject will undergo lateral DXA with VFA assessment, bone density assessment of each hip, radius and spine by DXA scan, bone structure assessment by HRpQCT of the distal radius and tibia, finite element assessment(µFEA), skin AGEs measurement, and blood collection to measure markers of bone formation and resorption.

ELIGIBILITY:
Inclusion Criteria:

Aim 1: Survey (Donors):

* Donated a kidney at one of the three participating sites.
* 10 or more years have passed since donation.
* Age ≥ 50 at time of study enrollment.

Aim 1: Survey (Controls):

* Subjects in the REP population.
* Medical records available for the five years preceding age at matching (age at donation).
* Matching will be based on: age, year of donation, sex, race/ethnicity, body mass index, comorbidity and selected risk factors (smoking, education level) status at year of donation

Aim 2: Skeletal health assessment (Donors and Controls):

* Subjects who have completed the survey
* Willing to come in for the in-person assessment

Exclusion Criteria:

Aim 1: Survey (Donors):

* Deceased
* Not willing to return the survey.

Aim 1: Survey (Controls):

* Deceased
* Not willing to return the survey
* History of the following conditions:

  * Diabetes mellitus, liver disease, kidney disease, nephrolithiasis, malabsorption syndrome, past history of non-traumatic fractures.

Aim 2: Skeletal health assessment (Donors and Controls):

* Subjects who did not participate in the survey
* Subjects not willing to come for the in-person evaluation.
* Women of childbearing potential.

Min Age: 50 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Living kidney donors who are more than 10 years post donation and who are 50 years of age or older at the time of study enrollment and matched controls.
Sampling Method: Non-Probability Sample
Enrollment: 4415 (Actual)
Dates: Start 2020-06-25 (Actual); Primary Completion 2023-08-04 (Actual); Study Completion 2023-08-04 (Actual)

PRIMARY OUTCOMES:
Evaluate bone health and bone fracture incidence in kidney donors and non-kidney donors | Baseline
  Measured by participant self-report response to survey about bone fractures and bone health survey
Changes in bone health after kidney donation | Day 1
  As indicated by comparisons between kidney donors and non-donors of dual-energy X-ray absorptiometry (DXA) measurements of bone mineral density at the lumbar spine (L1-L4), total hip and distal 1/3 of the forearm (GE Lunar) by DXA. Will be expressed as a T-score offset from expected peak bone mass as contained in the DXA scanner manufacturers' database.
Incidence of differences in bone architecture and strength after kidney donation | Day 1
  By comparisons of kidney donors and non-donors in measures of volumetric density and bone microarchitecture at the distal radius and tibia by high-resolution peripheral quantitative computed tomography (HR-pQCT). Bone strength will be evaluated using Image Processing Language (IPL) software to generate microfinite element (μFE) models from HR-pQCT imaging.
Incidence of changes in blood counts and blood chemistry measures after kidney donation | Day 1
  Based on variations between donors and non-donors in measures of complete blood count, serum electrolytes, Ca, Pi, creatinine, blood urea nitrogen and albumin.
Assess the correlations of bone biomarker and serum hormone concentrations with bone mineral density. | Day 1
  Based on comparison of bone and serum biomarkers in kidney donors and non-donors: (NTX; CTX; TRAcP5b; OC; BAP; P1NP; sclerostin assay); 1,25(OH)2D; 25(OH)D2 and 25(OH)D3; parathyroid hormone (PTH); fibroblast growth factor-23 (FGF23).
Assess the correlations of renal function with bone mineral health. | Day 1
  Renal function will be assessed by Measured Glomerular Filtration Rate (GFR), using the iothalamate short renal clearance technique, and by 24 hour urine collection to record the measures of creatinine clearance, urinary excretion of calcium, phosphorus, albumin and protein.

SECONDARY OUTCOMES:
Explore how vertebral Trabecular Bone Score (TBS) correlates with measures of bone health. | Day 1
  Trabecular bone score (TBS), a measure of bone quality, will be assessed from existing DXA images.
Evaluate Advanced Glycation Endproducts (AGEs) correlation to bone health parameters. | Day 1
  The AGEs Reader will measure the accumulations of AGEs in tissues in kidney donors and controls.

CONTACTS AND LOCATIONS:
Overall Officials: Rajiv Kumar, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

DOCUMENTS (1):
  • Informed Consent Form (2021-03-01): https://cdn.clinicaltrials.gov/large-docs/84/NCT04810884/ICF_000.pdf